CLINICAL TRIAL: NCT03203343
Title: Comparison of Inflammatory Stress Response Between Laparoscopic and Open Approach for Pediatric Inguinal Hernia Repair
Brief Title: Inflammatory Stress Response in Pediatric Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Miro Jukić, M.D., University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University hospital of Split
Record Dates: First submitted 2017-06-16; First posted 2017-06-29 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Inguinal Hernia, Indirect; Children, Only; Inflammatory Response; Surgery; Interleukin-6; Tumor Necrosis Factor Alpha; C Reactive Protein; White Blood Cell Count, Leukocytes
Keywords: Inguinal Hernia, Indirect; Children, Only; Inflammatory Response; Surgery; Interleukin-6; Tumor necrosis factor alpha; C reactive protein; Leukocytes
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIRS group (Active Comparator): Patients operated laparoscopically - PIRS technique
  Interventions: Procedure: Operation - PIRS
- Marcy group (Active Comparator): Patients operated by open modified Marcy technique
  Interventions: Procedure: Operation - MARCY

INTERVENTIONS:
Procedure: Operation - PIRS — Operation by its known design for PIRS group
  Arms: PIRS group
Procedure: Operation - MARCY — Operation by its known design for MARCY group
  Arms: Marcy group

SUMMARY:
Today there are various surgical techniques for inguinal hernia. In this study, investigators want to compare the ''PIRS'' operating technique laparoscopy and modified "Marcy" operating technique with open inguinal access. Investigators would compare both groups to find out witch one does the lesser inflammatory stress response on the organism.

DETAILED DESCRIPTION:
Inguinal hernia represents the protrusion of the abdominal cavity contents through the inguinal canal. Today there are various surgical techniques for inguinal hernia. In this study, investigators want to compare two standard methods that are regularly performed at the University hospital of Split at department of pediatric surgery. These are the ''PIRS'' operating technique laparoscopy and modified "Marcy" operating technique with open inguinal access. The choice of operating technique depends solely on the choice of a chosen pediatric surgeon. Given the fact that the child is indicated for an operation, regardless of participation in the study, there are no significant risks of participating in this study, except for possible but rare complications resulting from the peripheral venous blood draw (haematoma, soreness and pain). To carry out this study, the child should be taken (drawn) 3 peripheral venous blood samples (on day of operation, 24 hours after surgery and 6 days after surgery) from which the laboratory parameters are taken and counted (Leukocytes, C - Reactive Protein, Interleukin 6 and Tumor necrosis factor α).

Lab results would be compared between both groups to find out witch one does the lesser inflammatory stress response on the organism.

ELIGIBILITY:
Inclusion Criteria:

* male children with inguinal hernia at age of 3 to 7
* one-sided inguinal hernia

Exclusion Criteria:

* Female children
* recurrent hernia
* bilateral hernia
* age less than 3 y, more than 7 y
* any general inflammatory process, illness
* intraoperative complications which may interfere with inflammatory stress response

Ages: 3 Years to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male inguinal hernia
Enrollment: 32 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory stress response (IL6) | 3 measurements: preoperative, 24 hours after and 6 days after surgery
  measurement of IL6 in pg/mL (according to manufacturer), change of the value in three time frames like mentioned below
Change in inflammatory stress response (CRP) | 3 measurements: preoperative, 24 hours after and 6 days after surgery
  measurement of C - reactive protein in mg/L, change of the value in three time frames like mentioned below
Change in inflammatory stress response (TNF alpha) | 3 measurements: preoperative, 24 hours after and 6 days after surgery
  measurement of Tumor necrosis factor alpha in pg/mL (according to manufacturer), change of the value in three time frames like mentioned below
Change in inflammatory stress response (Leukocytes WBC) | 3 measurements: preoperative, 24 hours after and 6 days after surgery
  measurement of white blood cell count in 10^9/L, change of the value in three time frames like mentioned below

SECONDARY OUTCOMES:
Subjective pain assessment | 24 hours after and 6 days after surgery
  Visual analog pain scale
Subjective pain assessment | 6 days after surgery
  Visual analog pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Split, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Just investigators have insight in patient data, no such data (names and private data) would be written in the study for publishing

REFERENCES:
- [Derived] Jukic M, Pogorelic Z, Supe-Domic D, Jeroncic A. Comparison of inflammatory stress response between laparoscopic and open approach for pediatric inguinal hernia repair in children. Surg Endosc. 2019 Oct;33(10):3243-3250. doi: 10.1007/s00464-018-06611-y. Epub 2018 Dec 3. PMID 30511312